CLINICAL TRIAL: NCT04771260
Title: A Realist-informed Investigation of the Organisation and Delivery of Health and Social Care Services for People With Fibromyalgia Living in the UK
Brief Title: Understanding Health Services Delivery for Fibromyalgia
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 02/068/20
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Fibromyalgia; Fibromyalgia, Primary; Fibromyalgia, Secondary
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Case study #1: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #2: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #3: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #4: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #5: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #6: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #7: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #8: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #9: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.
- Case study #10: There will be no intervention. There will be 10 separate case studies, to identify how care for fibromyalgia is being delivered in each case study, and to identify models of care.

SUMMARY:
This research study aims to:

i) Explore and understand how health and social care for people with fibromyalgia living in the UK is organised and delivered.

ii) Identify models of practice to inform co-design of new care pathways for people with fibromyalgia living in the UK.

To do this, up to ten UK-based case studies will be conducted in total: at least one each in England, Scotland and Wales. Interviews will be conducted with approximately 10 participants per case study, for a total of 100 participant interviews. Qualitative observations (in-person or on-line) will be conducted with a similar number of people (total 100 participants). Online focus groups will also be carried out with approximately 6 to 8 participants per group (up to ten groups for a total 60-80 participants). Participants will include healthcare professionals (for example, doctors, nurses, allied health professionals), social care practitioners (for example, social prescribers), service delivery managers, commissioners and other individuals involved in the organisation and delivery of health and social care services for people with fibromyalgia living in the UK.

ELIGIBILITY:
Inclusion Criteria:

* NHS and/or non-NHS organisations in the UK providing health and social care to people with fibromyalgia.
* Health and social care professionals identifying and or providing support for people with fibromyalgia in one of the ten case studies.
* NHS/non-NHS staff influential in the organisation and/or delivery of health and social care to people with fibromyalgia in one of the ten case studies, for example, service managers, professional service leads, commissioners.

Exclusion Criteria:

* NHS/non-NHS organisations in the UK not providing health or social care to people with fibromyalgia.
* NHS/non-NHS staff who are not able to communicate sufficiently well in English to participate effectively.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include healthcare professionals (for example, doctors, nurses, allied health professionals), social care practitioners (for example, social prescribers), service delivery managers, commissioners and other individuals involved in the organisation and delivery of health and social care services for people with fibromyalgia living in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Model of care | By February 2022
  For each case study, how health and social care is being delivered will be the main outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2020-11-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04771260/Prot_000.pdf